CLINICAL TRIAL: NCT00903721
Title: Nasonex® Nasal Suspension 50 μg Long-term Designated Drug Use Investigation
Brief Title: Nasonex® Nasal Suspension 50 μg Long-term Designated Drug Use Investigation (Study P05876)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P05876
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Mometasone Furoate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with perennial allergic rhinitis
  Interventions: Drug: mometasone furoate
- 2: Patients with seasonal allergic rhinitis (including patients who also have perennial allergic rhinitis)
  Interventions: Drug: mometasone furoate

INTERVENTIONS:
Drug: mometasone furoate — Metered-dose spray type suspension containing 50 μg mometasone furoate per spray. 2 sprays per nostril twice daily (total daily dose 200 μg)
  Duration: up to 6 months
  Other Names: Nasonex® Nasal Suspension; Nasonex

SUMMARY:
The investigation will be conducted to define safety and efficacy under the conditions of post-marketing use of this drug in subjects with allergic rhinitis.

Post-marketing surveys are not considered applicable clinical trials and thus the results of this survey will not be posted at its conclusion. The results will be submitted to public health officials as required by applicable national and international laws.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are treated with Nasonex for perennial or seasonal allergic rhinitis.

Exclusion Criteria:

* Patients with an infection for which there is no effective antimicrobial drug or systemic fungal infection [symptoms may exacerbate]
* Patients with a history of hypersensitivity to any ingredient of this drug

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese patients with perennial allergic rhinitis and/or seasonal allergic rhinitis
Sampling Method: Non-Probability Sample
Enrollment: 3806 (Actual)
Dates: Start 2008-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Estimate the incidence of Adverse Drug Reactions (ADRs) | After 6 months of observation